CLINICAL TRIAL: NCT03230175
Title: A Multicenter, Open Label Phase 2 Pilot Trial of Subjects With Complex Non-healing Diabetic Foot Ulcers Treated With Standard Care Plus Cryopreserved Umbilical Cord Allograft (TTAX01)
Brief Title: Phase 2 Pilot Trial of Subjects With Complex Non-healing Diabetic Foot Ulcers Treated With Standard Care Plus Cryopreserved Umbilical Cord Allograft (TTAX01)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTCRNE-1501
Record Dates: First submitted 2017-07-19; First posted 2017-07-26 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Non-healing Wound; Non-healing Diabetic Foot Ulcer; Diabetic Foot Infection
MeSH Terms: interventions — Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TTAX01 plus standard care (Experimental): Eligible consenting subjects will undergo a baseline aggressive debridement in the operating room to remove infected and devitalized bone and soft tissue. A six week course of systemic antibiotics will be used to resolve baseline infection. TTAX01 will be applied to the debrided wound bed at baseline, and if healing is not evident, it will be applied again at 4 week intervals. At each weekly visit the wound will be further debrided as necessary.
  Interventions: Biological: TTAX01; Procedure: Surgical resection and debridement; Drug: Systemic antibiotics; Device: Off-loading

INTERVENTIONS:
Biological: TTAX01 — TTAX01 will be applied directly to the wound surface and retained with non-absorbable sutures. A single layer of the test article should cover the entire open surface of the wound. The material is to be applied once every 4 weeks unless the wound shows evidence of healing, in which case dosing is suspended; or, if the test article has been accidentally dislodged, it may be replaced at any time.
Procedure: Surgical resection and debridement — Perform surgical sharp debridement in the OR, to remove:
  * infectious agents and biofilms (purulence),
  * all debris, eschar, callus and macerated non-viable tissue from the wound base, and
  * dead (suprabasal epidermis), scarred (elevated/edematous) and necrotic/macerated tissue from the wound edge.
  Surgical Resection will be performed to remove as much of the necrotic bone detected by the radiographic evidence as is appropriate.
Drug: Systemic antibiotics — Six (6) weeks of systemic antibiotic therapy is required. A definitive therapy will be guided by the microbiological results based on bone biopsy.
Device: Off-loading — Provide off-loading device appropriate to the location of wound with full length boot or total contact cast

SUMMARY:
It is hypothesized that application of the human placental umbilical cord tissue TTAX01 to the surface of a well debrided, complex diabetic foot ulcer will, with concomitant management of infection, result in a higher proportion of wounds showing complete healing within 16 weeks of initiating therapy.

DETAILED DESCRIPTION:
The hypothesis under study is that one or more applications of TTAX01 to the wound surface of a well debrided, complex diabetic foot ulcer managed with appropriate antibiotic therapy will result in a higher probability of complete healing than would be expected from management with standard care alone. In this open label Phase 2 pilot trial, all subjects will receive the intervention over a maximum period of 16 weeks. Eligible consenting subjects will undergo a baseline aggressive debridement in the operating room to remove infected and devitalized bone and soft tissue. TTAX01 will be applied to the debrided wound bed at baseline, and if healing is not evident, it will be applied again at 4 week intervals. At each weekly visit the wound will be further debrided as necessary.

Consenting subjects who qualify for enrollment will undergo an aggressive surgical debridement at the baseline visit, including biopsies of bone for histology and microbiologic testing at the start and completion of debridement. Systemic antibiotics will be given empirically, with adjustments made on the basis of culture and sensitivity results. New or recurrent infections will be managed with additional debridement and adjustment or addition of appropriate systemic antibiotics. The test article, TTAX01, will be sutured to the debrided wound bed at baseline and again at 4 week intervals over the 16 week treatment period for wounds that do not show evidence of healing. For wounds that do show evidence of healing, additional applications of TTAX01 will be withheld, based on observations from retrospective case series.

Subjects whose wounds close prior to 16 weeks will move directly to a 2 week confirmation of closure period. Subjects whose wounds have not closed by the end of 16 weeks will exit the trial.

ELIGIBILITY:
Inclusion Criteria:

* The subject has signed the informed consent form
* The subject is male or female, at least 18 years of age inclusive at the date of Screening
* The subject has confirmed diagnosis of Type I or Type II diabetes
* The subject's index ulcer is located on the plantar surface, inter digital, heel, or lateral or medial surface of the foot
* The subject has an index ulcer with visible margins having an area ≥1.0 cm2 to ≤ 10.0 cm2 when measured by the electronic measuring device at Screening
* The subject's index ulcer extends beyond the dermis, into subcutaneous tissue with evidence of exposed bone, tendon, muscle and/or joint capsule
* The subject presents with history, signs or symptoms leading to a clinical suspicion of osteomyelitis in the opinion of the Investigator supported by positive Probe to Bone (PTB) and any of the following: radiographic (x-ray, Magnetic Resonance Imaging (MRI), or bone scan) or evidence of bone necrosis
* The subject has an Ankle Brachial Index ≥ 0.7 to ≤ 1.3 or TcPO2 ≥ 40 mmHg on the dorsum of the affected foot, or Great Toe Pressure ≥ 50 mmHg
* The subject is under the care of a physician for the management of Diabetes Mellitus

Exclusion Criteria:

* The subject's index ulcer is primarily located on the dorsal surface of the foot
* The subject's index ulcer can be addressed by primary closure through the completion of the initial or staged surgical procedure
* The subject has a glycated hemoglobin A1c (HbA1c) level of > 12%
* The subject has a serum albumin level ≤ 2.0 g/dL
* The subject has a white blood cell count < 2.0 x109/L, neutrophils < 1.0 x109/L, or platelets < 100 x109/L
* The subject has malignancy or a history of cancer, other than non-melanoma skin cancer, in five years before Screening
* The subject is pregnant
* The subject is a nursing mother
* The subject's index ulcer is over an active Charcot deformity
* The subject has had previous use of NEOX®, CLARIX®, or TTAX01 applied to the index ulcer
* Per Investigator's discretion the subject is not appropriate for inclusion in the trial, e.g., undergoing surgical treatments listed in the protocol or the subject currently has sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scheffer Tseng, MD, Study Chair — Chief Technology Officer
Locations (11):
- United States (11):
  - Banner University Medical Center, Phoenix, Arizona
  - UCLA Olive View, Sylmar, California
  - University of Miami, Miami, Florida
  - Village Podiatry Centers, Smyrna, Georgia
  - Rosalind Franklin University, North Chicago, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - St Luke's-Roosevelt Hospital Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - Carilion Clinic, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- TTAX01 Plus Standard Care: Eligible consenting subjects underwent a baseline aggressive debridement in the operating room to remove infected and devitalized bone and soft tissue. infection.
  TTAX01: TTAX01 was applied directly to the wound surface and retained with non-absorbable sutures. A single layer of the test article covered the entire open surface of the wound. The material was to be applied once every 4 weeks unless the wound shows evidence of healing, in which case dosing is suspended; or, if the test article has been accidentally dislodged, it may be replaced at any time.
  Surgical resection and debridement: Perform surgical sharp debridement in the OR, to remove:
  * infectious agents and biofilms (purulence),
  * all debris, eschar, callus and macerated non-viable tissue from the wound base, and
  * dead (suprabasal epidermis), scarred (elevated/edematous) and necrotic/macerated tissue from the wound edge.
  Surgical Resection will be performed to remove as much of the necrotic bone detected by the radiographic evidence as is appropriate.
  Systemic antibiotics: Six (6) weeks of systemic antibiotic therapy is required. A definitive therapy will be guided by the microbiological results based on bone biopsy.
  Off-loading: Provide off-loading device appropriate to the location of wound with full length boot or total contact cast
Period: Overall Study
Arm/Group | TTAX01 Plus Standard Care
Started | 32
Completed | 30
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- TTAX01 Plus Standard Care: Eligible consenting subjects underwent a baseline aggressive debridement in the operating room to remove infected and devitalized bone and soft tissue.
  TTAX01: TTAX01 was applied directly to the wound surface and retained with non-absorbable sutures. A single layer of the test article covered the entire open surface of the wound. The material was applied once every 4 weeks unless the wound shows evidence of healing, in which case dosing is suspended; or, if the test article has been accidentally dislodged, it may be replaced at any time.
  Surgical resection and debridement: Perform surgical sharp debridement in the OR, to remove:
  * infectious agents and biofilms (purulence),
  * all debris, eschar, callus and macerated non-viable tissue from the wound base, and
  * dead (suprabasal epidermis), scarred (elevated/edematous) and necrotic/macerated tissue from the wound edge.
  Surgical Resection will be performed to remove as much of the necrotic bone detected by the radiographic evidence as is appropriate.
  Systemic antibiotics: Six (6) weeks of systemic antibiotic therapy is required. A definitive therapy will be guided by the microbiological results based on bone biopsy.
  Off-loading: Provide off-loading device appropriate to the location of wound with full length boot or total contact cast
Arm/Group | TTAX01 Plus Standard Care
Number analyzed (Participants) | 32
Age, Customized [Number; unit: participants]
  < 65 years | 23
  > or = to 65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Alaskan Native/American Indian | 1
  Black/African American | 8
  White/Caucasian | 22
  Other, not specified | 1
Region of Enrollment [Number; unit: participants]
  United States | 32
Subject presents with history, signs or symptoms leading to a clinical suspicion of osteomyelitis [Count of Participants; unit: Participants] | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Complete Wound Healing
Description: Proportion of subjects with complete wound healing observed over the 16-week treatment period. Complete wound healing was defined as an initial observation of closure, followed by two confirmatory visits two weeks apart.
Time Frame: 16-weeks
Measure: Number; unit: participants
Groups:
- TTAX01 Plus Standard Care: Eligible consenting subjects underwent a baseline aggressive debridement in the operating room to remove infected and devitalized bone and soft tissue.
  TTAX01: TTAX01 was applied directly to the wound surface and retained with non-absorbable sutures. A single layer of the test article covered the entire open surface of the wound. The material was applied once every 4 weeks unless the wound shows evidence of healing, in which case dosing is suspended; or, if the test article has been accidentally dislodged, it was replaced at any time.
  Surgical resection and debridement: Performed surgical sharp debridement in the OR, to remove:
  * infectious agents and biofilms (purulence),
  * all debris, eschar, callus and macerated non-viable tissue from the wound base, and
  * dead (suprabasal epidermis), scarred (elevated/edematous) and necrotic/macerated tissue from the wound edge.
  Surgical Resection performed to remove as much of the necrotic bone detected by the radiographic evidence as is appropriate.
  Systemic antibiotics: Six (6) weeks of systemic antibiotic therapy was required. A definitive therapy was guided by the microbiological results based on bone biopsy.
  Off-loading: Provided off-loading device appropriate to the location of wound with full length boot or total contact cast
Arm/Group | TTAX01 Plus Standard Care
Number analyzed (Participants) | 32
participants | 16

2. Secondary Outcome: Time to Complete Wound Healing
Description: Time in number of days to complete wound closure over the 16 week treatment period, starting from enrollment to the time of the initial observation of wound closure
Time Frame: up to 16 weeks
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | TTAX01 Plus Standard Care
Number analyzed (Participants) | 32
weeks | 12.8 (4.3)

3. Secondary Outcome: Percent Change in Wound Surface Area
Description: Rate of wound closure, specifically percent change in the wound surface area (cm2) at each visit from baseline for assessing the rate of wound closure in area. Only percent change in wound surface area at week 16 reported.
Time Frame: at week 16
Measure: Mean (Full Range); unit: Percent Change
Arm/Group | TTAX01 Plus Standard Care
Number analyzed (Participants) | 32
Percent Change | 90.93 [84.54 to 95.31]

ADVERSE EVENTS:
Time Frame: The maximum time in the study for any subject was 21 weeks, with 1 week in screening and assuming wound healing occurs at week 16 followed by 2 weeks of observation for confirmation of closure, and a final exit visit 14 days later.
Description: An Adverse Event (AE) is any untoward medical occurrence temporally associated with the use of an investigational medicinal product, whether or not considered causally related to that product. An Serious Adverse Event is defined as any AE occurring at any dose that results in any of the following outcomes: death, life-threatening AE, requires hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect.
Arm/Group | TTAX01 Plus Standard Care
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 7/32
Other Adverse Events (participants affected / at risk) | 19/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TTAX01 Plus Standard Care (N=32)
Osteomyelitis (Infections and infestations) | 3 (3)
non-cardiac chest pain (General disorders) | 1 (1)
gastroparesis (Endocrine disorders) | 1 (1)
Bilateral Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
recurrent transient ischemic attack (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TTAX01 Plus Standard Care (N=32)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Diabetes mellitus inadequate control (Endocrine disorders) | 2 (2)
Diabetic Foot (Endocrine disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Osteomyelitis acute (Infections and infestations) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 2 (3)
Blister (Skin and subcutaneous tissue disorders) | 4 (6)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (7)
Skin maceration (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The one caveat is the lack of a control group. However, the study was designed to examine the safety and estimate the efficacy of TTAX01 plus standard care in achieving complete would closure of these complex non-healing diabetic foot ulcer with high risk factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT03230175/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT03230175/SAP_001.pdf